CLINICAL TRIAL: NCT01161316
Title: Phase-II, Randomized, Multicentre Pilot Study to Evaluate the Safety and Efficacy of the Treatment With mFOLFOX-6 Plus Cetuximab Versus Initial Treatment With mFOLFOX-6 Plus Cetuximab (for 8 Cycles), Followed by Maintenance With Cetuximab Alone as First-line Treatment in Patients With Metastatic Colorectal Cancer (mCRC) and Wild-type KRAS Tumours
Brief Title: Safety and Efficacy Study of mFOLFOX-6 Plus Cetuximab for 8 Cycles Followed by mFOLFOX-6 Plus Cetuximab or Single Agent Cetuximab as Maintenance Therapy in Patients With Metastatic Colorectal Cancer and WT KRAS Tumours
Acronym: MACRO-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-09-04; 2009-017194-38 (EudraCT Number)
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; wild-type KRAS tumours; cetuximab; mFOLFOX-6
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): mFOLFOX-6 + cetuximab until disease progression or early withdrawal.
  Interventions: Drug: mFOLFOX-6 + cetuximab until disease progression or early withdrawal.
- Experimental (Experimental): 8 cycles of mFOLFOX-6 + cetuximab, followed by cetuximab alone until disease progression or early withdrawal.
  Interventions: Drug: 8 cycles of mFOLFOX-6 + cetuximab, followed by cetuximab alone until disease progression or early withdrawal.

INTERVENTIONS:
Drug: mFOLFOX-6 + cetuximab until disease progression or early withdrawal. — Treatment regimen:
  mFOLFOX-6, day 1, every two weeks; OXALIPLATIN 85 mg/m2; FOLINIC ACID 400 mg/m2; 5-FU 400 mg/m2 IV bolus; 5-FU 2400 mg/m2 continuous infusion for 46 hours
  Cetuximab weekly. Cetuximab 400 mg/m2 the first time the treatment is administered; 250 mg/m2 for subsequent administrations.
  Arms: Control
Drug: 8 cycles of mFOLFOX-6 + cetuximab, followed by cetuximab alone until disease progression or early withdrawal. — Treatment regimen.
  mFOLFOX-6. day 1 every two weeks. OXALIPLATIN 85 mg/m2; FOLINIC ACID 400 mg/m2; 5-FU 400 mg/m2 IV bolus; 5-FU 2400 mg/m2 continuous infusion for 46 hours
  Cetuximab weekly. Cetuximab 400 mg/m2 the first time the treatment is administered; 250 mg/m2 for subsequent administrations.
  Arms: Experimental

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the combination of mFOLFOX-6 plus cetuximab for 8 cycles followed by mFOLFOX-6 plus cetuximab or single agent (s/a) cetuximab as maintenance therapy in patients (pts) with metastatic colorectal cancer (mCRC).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients of an age ≥ 18 years and < 71
* Patients with an ECOG performance status ≤ 2
* Confirmed histological diagnosis of colorectal carcinoma with metastatic disease and wild-type KRAS.
* Presence of at least one target lesion that is measurable one-dimensionally (not located in an irradiated region).
* Life expectancy greater than 12 weeks.
* First evidence of chemotherapy-naïve metastatic disease. Adjuvant chemotherapy is allowed if it has been more than 6 months since the treatment was finished and there have been no signs of disease progression, neither during treatment nor during the 6 months following its completion.
* Adequate medullar reserve:
* Absolute neutrophil count ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Haemoglobin ≥ 9 g/dL
* Adequate renal function: Creatinine clearance > 30 mL/min, calculated using the Cockroff-Gault formula, or a serum creatinine < 2 mg/dL or 177 umol/L
* An adequate liver function: ASAT (SGOT) and ALAT (SGPT) ≤ 2.5 x ULN (≤ 5 x ULN if there are liver metastases). Total bilirubin < 1.5 x ULN. Alkaline phosphatase ≤ 2.5 x ULN ( ≤ 5 x ULN in the case of liver metastases or ≤ 10 x ULN in the case of bone metastases)

Exclusion Criteria:

* To have received prior systemic treatment for the metastatic disease
* Diagnosis or suspicion of brain or leptomeningeal metastases
* Major surgery or radiotherapy (except for antalgic surgery that does not include measurable target lesions) during the 4 weeks prior to inclusion in the study.
* Previous administration of monoclonal antibodies, agents inhibiting EGFR signal transduction or EGFR-targeted treatment.
* Participation in another clinical trial with drugs within the previous 30 days.
* Neoplasm in the 2 years prior to entering the study, except for non-melanoma skin carcinoma or in situ cervix carcinoma.
* Evidence of previous acute hypersensitivity reaction of any degree to any of the treatment's components.
* Clinically relevant peripheral neuropathy.
* Signs and symptoms, at the moment of entering the study, of acute or subacute bowel obstruction.
* A history of an acute episode of ischemic heart disease (angina or acute myocardial infarction) within the previous 12 months or an elevated risk of heart failure decompensation or uncontrolled arrhythmia.
* Serious active infection, including active tuberculosis and HIV diagnosis.
* Chronic immunological or hormonal treatment, except for hormone replacement treatment at physiological doses.
* Known drug or alcohol abuse.
* Legal incapacity or limited legal capacity.
* Pregnancy or breastfeeding. Premenopausal women must have a negative pregnancy test in urine or blood before entering the trial. Patients and their partners must take contraceptive measures (hormonal, barrier, or abstinence) if the possibility of conception exists, during the study and for 3 months after the end of the treatment thereof.
* Any geographical or social circumstance or any medical or psychological alteration that, in the investigator's opinion, will not allow the patient to conclude the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2010-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 2010-2014

SECONDARY OUTCOMES:
overall survival | 2010-2014
rate of objective responses | 2010-2014
disease's resectability (R0) | 2010-2014
evaluate hypomagnesaemia as a predictive factor in the treatment's efficacy | 2010-2014
Adverse events | 2010-2014

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Aranda, Study Chair — Hospital Reina Sofia. Córdoba. Spain; Eduardo Díaz-Rubio, Study Chair — Hospital Clínico San Carlos. Madrid. Spain
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Benavides M, Diaz-Rubio E, Carrato A, Abad A, Guillen C, Garcia-Alfonso P, Gil S, Cano MT, Safont MJ, Gravalos C, Manzano JL, Sanchez A, Alcaide J, Lopez R, Massuti B, Sastre J, Martinez E, Escudero P, Mendez M, Aranda E. Tumour location and efficacy of first-line EGFR inhibitors in KRAS/RAS wild-type metastatic colorectal cancer: retrospective analyses of two phase II randomised Spanish TTD trials. ESMO Open. 2019 Dec 1;4(6):e000599. doi: 10.1136/esmoopen-2019-000599. eCollection 2019. PMID 31803504
- [Derived] Aranda E, Garcia-Alfonso P, Benavides M, Sanchez Ruiz A, Guillen-Ponce C, Safont MJ, Alcaide J, Gomez A, Lopez R, Manzano JL, Mendez Urena M, Sastre J, Rivera F, Gravalos C, Garcia T, Martin-Valades JI, Falco E, Navalon M, Gonzalez Flores E, Ma Garcia Tapiador A, Ma Lopez Munoz A, Barrajon E, Reboredo M, Garcia Teijido P, Viudez A, Cardenas N, Diaz-Rubio E; Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD). First-line mFOLFOX plus cetuximab followed by mFOLFOX plus cetuximab or single-agent cetuximab as maintenance therapy in patients with metastatic colorectal cancer: Phase II randomised MACRO2 TTD study. Eur J Cancer. 2018 Sep;101:263-272. doi: 10.1016/j.ejca.2018.06.024. Epub 2018 Jul 24. PMID 30054049
- See also: Related Info — http://www.ttdgroup.org